CLINICAL TRIAL: NCT05758922
Title: Randomized, Double Blind, Placebo Controlled, Multicenter, 12 Weeks Phase 2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AZ-3102 in Patients with GM2 Gangliosidosis or Niemann-Pick Type C Disease
Brief Title: Phase 2 Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AZ-3102 in Patients with GM2 Gangliosidosis or Niemann-Pick Type C Disease
Acronym: RAINBOW
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azafaros A.G. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZA-001-5A2-01
Record Dates: First submitted 2023-02-15; First posted 2023-03-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: GM2 Gangliosidosis; Niemann-Pick Disease, Type C
MeSH Terms: conditions — Gangliosidoses, GM2; Niemann-Pick Disease, Type C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participant will receive placebo once daily during the course of the study (12 weeks).
  Interventions: Drug: Placebo
- AZ-3102 (Dose 1) (Experimental): Participant will receive AZ-3102 (Dose 1) once daily during the course of the study (12 weeks) and the study extension (if applicable).
  Interventions: Drug: AZ-3102 (Dose 1)
- AZ-3102 (Dose 2) (Experimental): Participant will receive AZ-3102 (Dose 2) once daily during the course of the study (12 weeks) and the study extension (if applicable).
  Interventions: Drug: AZ-3102 (Dose 2)

INTERVENTIONS:
Drug: AZ-3102 (Dose 1) — Pharmaceutical form: capsule
  Route of administration: oral
  Arms: AZ-3102 (Dose 1)
Drug: Placebo — Pharmaceutical form: capsule
  Route of administration: oral
  Arms: Placebo
Drug: AZ-3102 (Dose 2) — Pharmaceutical form: capsule
  Route of administration: oral
  Arms: AZ-3102 (Dose 2)

SUMMARY:
This phase 2 is a randomized, double-blind, placebo controlled, 12 weeks study with daily oral administration of AZ-3102 aiming to evaluate the safety and pharmacokinetic (PK) profile in GM2 Gangliosidosis and Niemann-Pick type C disease (NP-C) patients. After approval by the country health authorities, a double-blind extension period was proposed to the patients who complete the 12-week study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged above 12 years old at informed consent signature.
* GM2 patients : Genetically and biochemically confirmed diagnosis of Tay-Sachs or Sandhoff disease.
* NP-C patients : Genetically confirmed diagnosis of NP-C.
* NP-C patients : Miglustat-naïve patients unwilling or unable to take miglustat, OR, patients who have discontinued miglustat because of confirmed safety/tolerability issues. Miglustat must have been discontinued at least 1 month prior to Baseline visit.
* Total SARA score ≥ 1 at Baseline.
* A male participant with a female partner of childbearing potential is eligible if he agrees to follow the contraceptive guidance.
* If a female participant is a WOCBP and is having a male partner, she must agree to follow the contraceptive guidance.
* Willing and able to complete protocol assessments.
* Parent and/or legal guardian is able to read, understand, and sign the informed consent. Where appropriate, assent will also be sought for patients who have not reached the age of majority or who are not able to sign the consent form.

Exclusion Criteria:

* Any abnormal conditions at baseline visit which, in the opinion of the PI; could interfere with study assessments (e.g., severe infection).
* History of medical conditions other than GM2 gangliosidosis/NP-C that, in the opinion of the PI; would confound scientific rigor or interpretation of results.
* Presence of another inherited neurologic disease.
* The dose of anti-epileptic treatment(s) was not stable and/or a new anti-epileptic treatment (drug or procedure) was prescribed during the last month before baseline.
* Total bilirubin >2 x ULN (isolated bilirubin >2 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
* Platelet count < 100 x 10^9/L.
* Presence of moderate or severe renal impairment.
* Prior participation in a clinical study with an investigational drug within 3 months prior to Baseline.
* Patient with a positive serum pregnancy test (tested only for women of childbearing potential) at baseline.
* Breast feeding ongoing at baseline or planned during the study.
* ECG with an average of triplicate QTcF interval > 440 msec.
* Received treatment with N-Acetyl-Leucine, gene therapy, stem cell transplantation, or with any other azasugars (iminosugars) compound with similar mechanism of action within 3 months before baseline (except for miglustat for which it is 1 month).
* Any known allergy to azasugars or any excipients.
* Evidence of suicidal ideation with intent (Type 4-5) on the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening. Only in patients judged by the PI cognitively capable to understand the concept of suicide.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety/tolerability: Incidence and severity of treatment emergent adverse events | Through study completion, up to Week 12
Assessment of pharmacokinetic (PK) parameters in plasma: Cmax | Through study completion, up to Week 12
Assessment of PK parameters in plasma: Tmax | Through study completion, up to Week 12
Assessment of PK parameters in plasma: AUC0-24h | Concentration versus time curve calculated from time 0 to 24 hours (AUC0-24h)

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Hospital Pequeno Principe, Curitiba
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Instituto Nacional de Saúde da Mulher, da Criança e do Adolescente Fernandes Figueira, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No